CLINICAL TRIAL: NCT07112339
Title: EFFectiveness of Once-weekly Insulin ICodec Versus Once-daily Basal Insulin Analogues in an Insulin-naïve Type 2 diabEtes Population in Real-world cliNical pracTice- The EFFICIENT Pragmatic Study Effectiveness of Insulin Icodec in Real-world Clinical Practice
Brief Title: A Research Study to See How Well Weekly Insulin Icodec Maintains Blood Sugar Levels Compared to Daily Basal Insulins in Adults With Type 2 Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-7727; U1111-1302-4943 (Other: World Health Organization (WHO)); 2024-520068-32 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin icodec (Experimental): Participants will receive subcutaneous (s.c) injection of once weekly insulin icodec.
  Interventions: Drug: Insulin icodec
- Basal insulin analogues (Active Comparator): Participants will receive once daily s.c. injection of basal insulin analogues.
  Interventions: Drug: Basal insulin analogues

INTERVENTIONS:
Drug: Insulin icodec — Insulin icodec will be administered as subcutaneous injection.
  Arms: Insulin icodec
Drug: Basal insulin analogues — Basal insulin analogues will be administered as subcutaneous injection.
  Arms: Basal insulin analogues

SUMMARY:
This study compares insulin icodec, taken once a week, with other basal insulins, taken once a day, in people with type 2 diabetes.The purpose of this study is to see how well the approved injectable weekly insulin icodec maintains blood sugar levels when compared to approved and available daily injectable basal insulins in people with type 2 diabetes. The participants will either be prescribed weekly insulin icodec or a daily basal insulin (insulin glargine, insulin detemir or insulin degludec) based on current standards for the treatment of type 2 diabetes. The study will last for about 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2D greater than or equal to (≥) 180 days prior to the day of screening.
* Treatment with any of the following non-insulin glucose-lowering medication(s) or combination regimen(s) at the time of screening:

Metformin, Sulfonylureas, Meglitinides (glinides), dipeptidyl peptidase-4 (DPP-4) inhibitors, sodium-glucose cotransporter-2 (SGLT2) inhibitors, Thiazolidinediones, Alpha-glucosidase inhibitors, Oral combination products (for the allowed individual oral antidiabetic drugs), Oral or injectable glucagon-like peptide-1 (GLP-1) receptor agonists and Injectable dual glucose-dependent insulinotropic polypeptides (GIP) and GLP-1 receptor agonist.

* Need of intensification with basal insulin, as indicated at the discretion of the investigator.
* Recorded HbA1c value ≥7% within the last 90 days prior to randomization.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Previous participation in this study. Participation is defined as signed informed consent.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive method.
* Participation (i.e., received any study intervention) in any interventional clinical study within 90 days before screening.
* Any disorder which in the investigator's opinion might jeopardize participant's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline week 0 to week 52
  Measured as %-point.

SECONDARY OUTCOMES:
Adelphi Adherence Questionnaire (ADAQ©) | At week 52
  Measured as Score. The ADAQ© score is calculated as the mean of 11 individual items, each rated on a scale from 0 to 4. To obtain the mean score, at least 8 of these items must be answered. A lower score indicates greater adherence.
Change in Diabetes Treatment Satisfaction Questionnaire- status version(DTSQs) total treatment satisfaction | From baseline week 0 to week 52
  Measured as Score of 0-36. DTSQs score ranges from 0 to 36, based on 6 items that are each rated on a scale of 0 to 6. A higher score reflects greater satisfaction with the treatment received.
Treatment Related Impact Measure for Diabetes (TRIM-D) compliance domain | At week 52
  Measured as Score of 4-20.The score ranges from 4 to 20, based on 4 items rated on a scale of 1 to 5. This score is then transformed to a 0-100 scale, where higher scores indicate better compliance.
Treatment Related Impact Measure for Diabetes (TRIM-D) treatment burden domain | At week 52
  Measured as Score of 6-30. The score ranges from 6 to 30, derived from 6 items each rated on a scale of 1 to 5. This score is then transformed to a 0-100 scale, where higher scores indicate less treatment burden.
Number of severe hypoglycaemic episodes (level 3) | From baseline week 0 to week 52
  Measured as Number of episodes.
Mean weekly basal insulin dose | From week 50 to week 52
  Measures in Units.
Participant achieved individualised HbA1c target | At week 52
  Reported as Yes or No.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (75):
- Canada (39):
  - Centricity Research Calgary Endocrinology, Calgary, Alberta
  - Alta Clinical Research at Hermitage Medicentre, Edmonton, Alberta
  - Fraser Clinical Trials Inc., New Westminster, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Centricity Research Brampton Endocrinology, Brampton, Ontario
  - Centricity Clinical Research Burlington, Burlington, Ontario
  - Centricity Research Vaughn Endocrinology, Concord, Ontario
  - Medical Trust Clinics, Inc., Courtice, Ontario
  - Centricity Research Etobicoke Endocrinology, Etobicoke, Ontario
  - Janik Research, Greater Sudbury, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - St. Josephs Health Care, London, Ontario
  - Western Univ. Cnt for Studies in Fam Med, London, Ontario
  - Malton Medical Clinic, Mississauga, Ontario
  - Centricity Research Ottawa LMC, Nepean, Ontario
  - The Ottawa Hospital_Riverside, Ottawa, Ontario
  - Bluewater Clin Res Group Inc, Sarnia, Ontario
  - Sewa Ram Singal Medicine Professional Corp, Toronto, Ontario
  - Centricity Research Toronto, Toronto, Ontario
  - Centricity Research Toronto Manna Multispec, Toronto, Ontario
  - Diex Recherche Joliette, Joliette, Quebec
  - Alpha Recherche Clinique - Clinique de Levis, Lévis, Quebec
  - Centricity Research Mirabel, Mirabel, Quebec
  - Centre hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Applied Medical Informatics Research, Montreal, Quebec
  - Clinique Endocrinologie OASIS., Montreal, Quebec
  - Centricity Res Pointe-Claire, Pointe-Claire, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Centre de Recherche Saint-Louis, Sherbrooke, Quebec
  - Ctr de Med Metab de Lanaudiere, Terrebonne, Quebec
  - Diex Recherche Trois-Rivieres, Trois-Rivières, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
  - Recherche Clinique Sigma Inc., Québec
  - Diex Recherche Quebec Inc., Québec
  - Centre de Recherche Saint-Louis, Québec
  - Alpha Recherche Clinique - Lebourgneuf, Québec
- Germany (23):
  - Versidas - Diabetologikum Amberg, Amberg, Bavaria
  - Diabetespraxis Mergentheim, Bad Mergentheim
  - Praxis Dr. Stephan Scharla, Bad Reichenhall
  - Medizinisches Versorgungszentrum Am Bahnhof Spandau GbR, Berlin
  - Studiengesellschaft Dres. Könemann/Steinmann GbR, Bünde
  - Diabetologische Schwerpunktpraxis Daaden, Daaden
  - Diabeteszentrum-Do Dres. K U. Ch. Busch GbR, Dortmund
  - Studienzentrum Dr. Faulmann GbR Dresden, Dresden
  - MVZ Hausärzte Großenbaum GmbH Duisburg, Duisburg
  - Praxis für Diabetologie, Angiologie und Innere Medizin Eisenach, Eisenach
  - MVZ Contilia GmbH, Essen
  - Praxis am Markt Dr. Becker, Essen
  - MVZ im Altstadt-Carree Fulda GmbH - Zentrum für klinische Studien, Fulda
  - Diabetes-Zentrum-Wilhelmsburg GbR, Hamburg
  - Mesut Durmaz, Hof, Hof
  - Praxisgemeinschaft Jerichow, Jerichow
  - Familienmedizinisches Zentrum Radowsky, Leipzig
  - Praxis Am Oberen Tor - Dr. Simon-Wagner, Lichtenfels
  - Diabeteszentrum Ludwigsburg, Ludwigsburg
  - Institut für Diabetesforschung Osnabrück, Osnabrück
  - ceda - Centrum für Diabetologie und Allgemeinmedizin Pohlheim, Pohlheim
  - Hegau-Bodensee-Klinikum Singen, Singen
  - Dr. Schmidt-Reinwald Astrid, Trier, Trier
- Italy (13):
  - A.O.U. Consorziale Policlinico di Bari, Bari, BA
  - AOU Vanvitelli - DAI Medicina Interna, Geriatria e Neurologia - U.O.C. Endocrinologia e Malattie del Metabolismo, Napoli, Campania
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Centro malattie endocrine e metaboliche, Rome, Lazio
  - DAI Scienze Mediche - UOC Endocrinologia, Messina, Sicily
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone - Presidio Villa Belmonte, Palermo, Sicily
  - AST Fermo - Ospedale Murri - Unità Operativa di Diabetologia e Endocrinologia, Fermo, The Marches
  - Azienda Ospedaliero Universitaria Careggi - Diabetologia e malattie del metabolismo, Florence, Tuscany
  - Azienda Ospedaliera di Perugia;Ospedale S. Maria della Misericordia, Perugia, Umbria
  - Policlinico Mater Domini Università di Catanzaro, Catanzaro
  - Università degli studi G. D'Annunzio Chieti Pescara - CAST, Chieti Scalo
  - Azienda Ospedaliera Luigi Sacco, Milan
  - AUSL Romagna - Medicine Specialistiche Ravenna - UO Servizio di Diabetologia di Ravenna, Ravenna
  - Azienda Ospealiero Universitaria Policlinico Umberto I, Roma

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com